CLINICAL TRIAL: NCT04800510
Title: Iterative Design of Custom Dynamic Orthoses and Comprehensive Design of Musculoskeletal Model
Brief Title: Iterative Design of Custom Dynamic Orthoses
Acronym: PRMRP-Norms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jason Wilken, Associate Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 202002131; CDMRP-PR172087 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2023-12

CONDITIONS: Adult ALL; Healthy
Keywords: Gait Analysis; Ankle Foot Orthosis; Carbon Fiber; Biomechanics
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: All participants will use three generic sized carbon fiber custom dynamic orthoses (CDOs). Each CDO will differ from the others in design and will be labeled as CDO-A, CDO-B and CDO-C. Participants will be randomly assigned to one of six CDO testing sequences (ABC, ACB, BCA, BAC, CAB, CBA) to prevent testing order from influencing study results.
Who Masked: Participant
Masking Description: Participants will be blinded to the different design variations of each device, and will only be introduced to each device as CDO-A, CDO-B or CDO-C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- NoCDO, CDOA, CDOB, CDOC (Experimental): Participants will be evaluated without a CDO, then with CDOA, then with CDOB, then with CDOC.
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- NoCDO, CDOA, CDOC, CDOB (Experimental): Participants will be evaluated without a CDO, then with CDOA, then with CDOC, then with CDOB.
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- NoCDO, CDOB, CDOA, CDOC (Experimental): Participants will be evaluated without a CDO, then with CDOB, then with CDOA, then with CDOC.
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- NoCDO, CDOB, CDOC, CDOA (Experimental): Participants will be evaluated without a CDO, then with CDOB, then with CDOC, then with CDOA.
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- NoCDO, CDOC, CDOA, CDOB (Experimental): Participants will be evaluated without a CDO, then with CDOC, then with CDOA, then with CDOB.
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- NoCDO, CDOC, CDOB, CDOA (Experimental): Participants will be evaluated without a CDO, then with CDOC, then with CDOB, then with CDOA.
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)

INTERVENTIONS:
Device: Carbon Fiber Custom Dynamic Orthosis (CDO) — The CDO will consist of a semi-rigid foot plate, a posterior carbon fiber strut, and a proximal cuff below the knee.
  Other Names: Ankle Foot Orthosis

SUMMARY:
The proposed study evaluates the effect of carbon fiber brace design on forces across the ankle joint. It is expected that carbon fiber braces can be designed to reduce forces in the ankle. In this study, brace geometry will be varied to determine how these changes influence the forces experienced by ankle cartilage. The purpose of this study is to refine a pre-existing musculoskeletal model and finalize the procedures for inputting multiple data sources into the model to evaluate ankle articular contact stresses.

DETAILED DESCRIPTION:
The purpose of this study is to refine a pre-existing musculoskeletal model and finalize the procedures for inputting multiple data sources into the model to evaluate ankle articular contact stresses.

Healthy adult participants will complete testing using three generic sized carbon fiber custom dynamic orthoses (CDOs) and with no CDO. Participants will be blinded to the design variation of each device and will only know them as CDO-A, CDO-B, or CDO-C. Testing will be completed under 4 conditions: No-CDO, CDO-A, CDO-B, CDO-C, with each bracing condition (A/B/C) representing a CDO design variant. Physical performance measures will incorporate tests of agility, speed, and lower limb power to ensure that changes to device design do not negatively affect physical function. Questionnaires will be used to evaluate participants' current and desired activity level, pain with and without CDO use, satisfaction with the devices, perception of comfort and smoothness between devices, and preference between CDOs. Semi-structured interviews will be completed to fully capture the participant's perspective. Lower limb forces and motion will be assessed using a computerized motion capture system and force plates in the floor. Forces between the foot and CDO will be measured using force sensing insoles, and muscle activity data will be collected using surface electromyography. Devices will be mechanically tested, and participant demographic and anthropometric data will be recorded.

The information obtained from this study will help refine the musculoskeletal model data input methods to be used in future studies. The knowledge that will be gained from this investigation has the potential to substantially improve the long-term efficacy and efficiency of the musculoskeletal model and help improve ankle foot orthosis

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 50
* Shoe size between women's 8 and 13.5 or men's 6.5 and 12
* Healthy individuals without a current complaint of lower extremity pain, spine pain, or medical or neuromusculoskeletal disorders that have limited participation in work or exercise in the last 6 months
* Full active range of motion of the bilateral lower extremities and spine
* Ability to hop without pain
* Ability to perform a full squat without pain
* Ability to read and write in English and provide written informed consent

Exclusion Criteria:

* Diagnosed moderate or severe brain injury
* Prior lower extremity injury resulting in surgery or limiting function for greater than 6 weeks
* Diagnosis of a physical or psychological condition that would preclude testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
* Visual or hearing impairment that would interfere with instructions given during testing
* Require an assistive device
* Wounds to the foot or calf that would prevent CDO use
* BMI greater than 35
* Pregnancy - Per participant self-report. Due to the expected small number of pregnant individuals and resulting inability to account for its effect on resulting outcomes, participants will be withdrawn from the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NoCDO, CDOA, CDOB, CDOC | NoCDO, CDOA, CDOC, CDOB | NoCDO, CDOB, CDOA, CDOC | NoCDO, CDOB, CDOC, CDOA | NoCDO, CDOC, CDOA, CDOB | NoCDO, CDOC, CDOB, CDOA
Started | 0 | 4 | 1 | 1 | 2 | 1
Completed | 0 | 4 | 1 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No study participants were randomized to testing order NoCDO, CDOA, CDOB, CDOC
Groups:
- Total: Total of all reporting groups
Arm/Group | NoCDO, CDOA, CDOB, CDOC | NoCDO, CDOA, CDOC, CDOB | NoCDO, CDOB, CDOA, CDOC | NoCDO, CDOB, CDOC, CDOA | NoCDO, CDOC, CDOA, CDOB | NoCDO, CDOC, CDOB, CDOA | Total
Number analyzed (Participants) | 0 | 4 | 1 | 1 | 2 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 21.8 (2.1) | 23.0 (0.0) | 22.0 (0.0) | 22.5 (0.7) | 19.0 (0.0) | 21.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 0 | 0 | 1 | 4
  Male | 0 | 1 | 1 | 1 | 2 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 4 | 1 | 1 | 2 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 4 | 1 | 0 | 2 | 0 | 7
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Joint Contact Stress-Time Exposure
Description: Joint contact stress-time exposure (MPA-s/gait cycle) will be estimated using a participant specific musculoskeletal model. The model included surface geometry of each participants tibia and talus. Contact stress -time exposure, measured in MPa-s, was calculated at 13 points across the gait cycle. Higher values indicate greater contact stress-time exposure.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: MPa-s/gait cycle
Groups:
- NoCDO: Participants completed testing without an orthosis.
- CDOA: Participants completed testing in a carbon fiber custom dynamic orthosis: CDOA, a moderate stiffness PhatBrace (Bio-Mechanical Composites, Des Moines, IA)
- CDOB: Participants completed testing in a carbon fiber custom dynamic orthosis: CDOB, a firm stiffness PhatBrace (Bio-Mechanical Composites, Des Moines, IA)
- CDOC: Participants completed testing in a carbon fiber custom dynamic orthosis: CDOC, the Malleo-Lok (Bio-Mechanical Composites, Des Moines, IA)
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
MPa-s/gait cycle | 3.9 (2.9) | 3.5 (2.7) | 4.1 (2.9) | 2.7 (0.6)

2. Secondary Outcome: Ankle Range of Motion
Description: Peak dorsiflexion angle (degrees) during gait.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
degrees | 17.8 (3.3) | 16.0 (3.4) | 16.3 (2.8) | 15.5 (3.6)

3. Secondary Outcome: Peak Ankle Moment
Description: Peak ankle moment (Nm/kg) during gait.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
Nm/kg | 1.5 (0.1) | 1.5 (0.1) | 1.5 (0.1) | 1.4 (0.1)

4. Secondary Outcome: Peak Ankle Power
Description: Peak ankle power (W/kg) during gait.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
W/kg | 2.9 (0.8) | 1.8 (0.3) | 1.6 (0.3) | 2.4 (0.4)

5. Secondary Outcome: Plantar Force (Total Foot)
Description: Force data (N) collected across the total foot measured between the foot and orthosis during gait.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
N/kg | 406.5 (64.7) | 415.1 (80.5) | 428.6 (82.2) | 424.7 (83.3)

6. Secondary Outcome: Plantar Force (Forefoot)
Description: Force data (N) collected across the forefoot (distal 40% of insole) measured between the foot and orthosis during gait.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
N/kg | 199.0 (42.6) | 165.7 (47.3) | 135.2 (42.0) | 149.9 (50.4)

7. Secondary Outcome: Plantar Force (Midfoot)
Description: Force data (N) collected across the midfoot (middle 30% of insole) measured between the foot and orthosis during gait.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
N/kg | 65.4 (19.1) | 83.5 (21.4) | 81.6 (33.8) | 89.9 (32.9)

8. Secondary Outcome: Plantar Force (Hindfoot)
Description: Force data (N) collected across the hindfoot (proximal 30% of insole) measured between the foot and orthosis during gait.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
N/kg | 142.0 (39.5) | 165.9 (47.2) | 211.8 (75.6) | 184.9 (62.5)

9. Secondary Outcome: Four Square Step Test (4SST)
Description: The 4SST (s) is a standardized timed test of balance and agility.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
seconds | 5.5 (1.7) | 6.1 (1.5) | 6.1 (1.7) | 5.8 (1.5)

10. Secondary Outcome: Sit to Stand 5 Times (STS5)
Description: STS5 (s) is a well-established timed measure of lower limb muscle strength and power. Participants are instructed to stand up and sit down 5 times as fast as possible.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
seconds | 7.0 (1.8) | 7.7 (1.7) | 7.4 (1.7) | 7.2 (1.5)

11. Secondary Outcome: Numerical Pain Rating Scale
Description: Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable.
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
score on a scale | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

12. Secondary Outcome: The Orthotics Prosthetics Users' Survey (OPUS)
Description: Satisfaction with device will be assessed using the Orthotics Prosthetics Users' Survey Satisfaction With Device Score. The survey asks users to indicate how much they agree with each statement on a scale from - Strongly Agree (5) to Strongly Disagree (0) with a Don't Know/Not Applicable option. The average score across all questions was calculated and reported, larger scores indicate a better outcome associated with that device. The maximum possible score is a 5 and the minimum possible score is a 0.
Time Frame: Baseline
Population: The OPUS questionnaire does not apply to none-braced conditions, as such each of the study participants completed the questionnaire in all braced conditions: CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9
score on a scale | 3.5 (0.4) | 3.6 (0.3) | 4.0 (0.4)

13. Secondary Outcome: Soleus Muscle Force (N)
Description: Peak Soleus muscle forces (N) will be estimated using an Opensim model
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: N
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
N | 1813.0 (505.7) | 1250.2 (596.5) | 1106.6 (358.2) | 1466.3 (394.3)

14. Secondary Outcome: Gastrocnemius Muscle Force (N)
Description: Peak Gastrocnemius muscle forces (N) will be estimated using an OpenSim model
Time Frame: Baseline
Population: Each of the study participants completed testing in all conditions: NoCDO, CDOA, CDOB, CDOC
Measure: Mean (Standard Deviation); unit: N
Arm/Group | NoCDO | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9 | 9
N | 1232.6 (321.7) | 1333.9 (425.9) | 1262.3 (394.6) | 1210.5 (240.2)

15. Secondary Outcome: Modified Socket Comfort Score (Comfort)
Description: Comfort scores range from 0 = most uncomfortable to 10 = most comfortable.
Time Frame: Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9
score on a scale | 6.6 (2.2) | 6.8 (1.9) | 8.0 (1.9)

16. Secondary Outcome: Modified Socket Comfort Score (Smoothness)
Description: Comfort scores range from 0 = least smooth to 10 = most smooth.
Time Frame: Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CDOA | CDOB | CDOC
Number analyzed (Participants) | 9 | 9 | 9
score on a scale | 6.6 (2.1) | 6.9 (2.3) | 8.3 (1.3)

17. Other Pre Specified Outcome: Participant Device Preference
Description: The participant will rank order their preference for their standard of care device (if applicable), No Device, CDO-A, CDO-B, CDO-C on a questionnaire.
Time Frame: Baseline
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Semi-Structured Interview
Description: Semi-structured interviews will also be used to fully capture the patients' perspectives, experience, and opinions associated with the device options they experienced as part of the study.
Time Frame: Baseline
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Center of Pressure Velocity Timing
Description: Timing of peak center of pressure velocity (percent stance) during gait.
Time Frame: Baseline
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Center of Pressure Velocity Magnitude
Description: Magnitude of peak center of pressure velocity (m/s) during gait.
Time Frame: Baseline
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Soleus Muscle Activity (Electromyography)
Description: Electromyography (EMG, % Maximum) of the Soleus during gait.
Time Frame: Baseline
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Rectus Femoris Muscle Activity (Electromyography)
Description: Electromyography (EMG, % Maximum) of the Rectus Femoris during gait.
Time Frame: Baseline
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Vastus Medialis Muscle Activity (Electromyography)
Description: Electromyography (EMG, % Maximum) of the Vastus Medialis during gait.
Time Frame: Baseline
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Medial Gastrocnemius Muscle Activity (Electromyography)
Description: Electromyography (EMG, % Maximum) of the Medial Gastrocnemius during gait.
Time Frame: Baseline
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Tibialis Anterior Muscle Activity (Electromyography)
Description: Electromyography (EMG, % Maximum) of the Tibialis Anterior during gait.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study participants were asked to indicate any adverse events throughout the duration of the study visit. After completion of the study visit participants were also asked to call or email the research team if any adverse events related to the study occurred after the study visit (up to ~12 months after the visit).
Description: No study participants were randomized to testing order NoCDO, CDOA, CDOB, CDOC so no participants in that group were at risk for Serious Adverse Events, All-Cause Mortality, or Other Adverse Events
Groups:
- NoCDO: Participants will be evaluated without a CDO.
- CDOA: Participants will be evaluated with CDOA.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a semi-rigid foot plate, a posterior carbon fiber strut, and a proximal cuff below the knee.
- CDOB: Participants will be evaluated with CDOB.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a semi-rigid foot plate, a posterior carbon fiber strut, and a proximal cuff below the knee.
- CDOC: Participants will be evaluated with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a semi-rigid foot plate, a posterior carbon fiber strut, and a proximal cuff below the knee.
Arm/Group | NoCDO | CDOA | CDOB | CDOC
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT04800510/Prot_SAP_001.pdf